CLINICAL TRIAL: NCT07232199
Title: Clinical Investigation of Sensovisc Sterile Sodium Hyaluronate Gel in the Hip Joint
Brief Title: Clinical Investigation of Sensovisc Sterile Sodium Hyaluronate Gel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: İstem Medikal Tıbbi Cihaz ve Sanayi Ticaret Anonim Şirketi (Unknown)
Responsible Party: Principal Investigator, Emre Adıgüzel, Prof. MD, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkentHayriyesimsek03
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis
Keywords: viscosupplementation; hip osteoarthritis; hyaluronic acid; intraarticular injection; Sensovisc
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensovisc® (Experimental): Other Names: Hyaluronic Acid Gel,Intra-articular injection,Sodium Hyaluronate Injectable Sterile Sodium Hyaluronate Gel
  Interventions: Device: SV-3-75: Sterile Sodium Hyaluronate Gel-3 mL Prefilled Syringe (2.5%)

INTERVENTIONS:
Device: SV-3-75: Sterile Sodium Hyaluronate Gel-3 mL Prefilled Syringe (2.5%) — Sensovisc is used to reduce osteoarthritis related pain in the joints by supporting synovial fluid by intra-articular injection and allowing the synovial fluid to restore its viscoelastic properties. It increases the joint mobility by reducing or eliminating the pain. It will be injected in hip joint in this investigation. The injection will be administered under fluoroscopic and ultrasound guidance.

SUMMARY:
This clinical investigation aims to investigate the safety and performance of Sensovisc.Sensovisc is used to reduce osteoarthritis related pain in the joints by supporting synovial fluid by intra-articular injection and allowing the synovial fluid to restore its viscoelastic properties. It increases the joint mobility by reducing or eliminating the pain.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most prevalent chronic arthritis and a leading cause of pain and disability among adults. OA is a degenerative joint disease characterized by chronic inflammation, cartilage degradation and erosion of underlying bone in the affected joints, predominantly affects knees, significantly impacting patient mobility and quality of life. • Although there are currently no approved disease-modifying OA drugs (DMOADs), nonpharmacologic interventions, such as physical therapy and weight management, and pharmaceutical approaches are available to reduce or revise joint damage and inflammation.• Among various therapeutic interventions, intra-articular hyaluronic acid (HA) injections have emerged as an alternative promising treatment. Emerging evidence suggests that HA may exert chondroprotective effects by enhancing synovial fluid viscosity, improving joint lubrication, and mitigating inflammatory processes, thereby potentially decelerating disease progression and preserving cartilage integrity.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients who have unilateral and/or bilateral hip pain for more than 3 months and meet the diagnosis of coxarthrosis according to ACR criteria
* 40 mm above the pain level determined by the Visual Analogue Scale (VAS) during rest for at least 15 days in the month before starting the study (for paracetamol and oral NSAIDs, taking into account the half-life of the drug).
* Diagnosis of hip osteoarthritis with Stage II or III according to the Kellgren and Lawrence (KL) classification, as determined by x-rays taken in the last 12 months
* Ambulating with or without support
* Having the mental ability to express pain scores
* Signing the informed consent form indicating consent to participate in the study

Exclusion Criteria:

* Radiological Kellgren-Lawrence (K&L) stage I or IV
* Other non-degenerative causes of hip pain
* septic arthritis
* Avascular necrosis,
* Femoroacetabular impingement syndrome,
* Trochanteric bursitis
* Having a history of lower extremity fracture/surgery within the last 6 months
* Pregnancy, breastfeeding, pregnancy plan
* Morbidly obese patients (BMI>40),
* Patients with unstable medical conditions (liver or kidney failure, lung/heart disease, tumor, HIV, etc.)
* Known central nervous system and/or peripheral nervous system disease
* When fluoroscopy guided injection is contraindicated:

  * pregnancy,
  * contrast material allergy,
  * local anesthetic allergy,
  * Having conditions such as coagulopathy
* Related to Treatment

  * Corticosteroid injection into the target joint within the last 1 month before the first injection
  * Hyaluronan injection into the target joint within the last 6 months before the first injection
  * Arthroscopy or surgery on the target joint within the last 6 months before the first injection
* Those who use blood thinners (warfarin compounds and heparin) or have bleeding problems
* Contraindications for SENSOVISC: Hypersensitivity to product ingredients, systemic infection, presence of local infection on the buttocks, infection or skin disease at the injection site or joint area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
Change in Visual Analogue Scale (VAS) score from baseline at 6 weeks | 6 weeks after the injection
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
Change in Visual Analogue Scale (VAS) score from baseline at 6 months | 6 months after the injection
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
WOMAC Osteoarthritis Index | Baseline
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Change in WOMAC Osteoarthritis Score from baseline at 6 weeks | 6 weeks after the injection
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Change in WOMAC Osteoarthritis Score from baseline at 6 months | 6 months after the injection
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Harris Hip Score (HHS) | Baseline
  It is a clinician-administered tool used to assess hip pain, function, deformity, and range of motion, with a total score ranging from 0 to 100 (higher scores indicate better function). Scores are categorized as excellent (90-100), good (80-89), fair (70-79), and poor (<70). The HHS will be used to evaluate hip function before and after the intervention.
Change in Harris Hip Score (HHS) from baseline at 6 weeks | 6 weeks after last injection
  It is a clinician-administered tool used to assess hip pain, function, deformity, and range of motion, with a total score ranging from 0 to 100 (higher scores indicate better function). Scores are categorized as excellent (90-100), good (80-89), fair (70-79), and poor (<70). The HHS will be used to evaluate hip function before and after the intervention.
Change in Harris Hip Score (HHS) from baseline at 6 weeks | 6 months after last injection
  It is a clinician-administered tool used to assess hip pain, function, deformity, and range of motion, with a total score ranging from 0 to 100 (higher scores indicate better function). Scores are categorized as excellent (90-100), good (80-89), fair (70-79), and poor (<70). The HHS will be used to evaluate hip function before and after the intervention.